CLINICAL TRIAL: NCT07310381
Title: Vagus Nerve Stimulation (VNS) Electroencephalogram (EEG) Protocol Supplement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Wallace Austelle, Clinical Assistant Professor, Department of Psychiatry & Behavioral Sciences, Stanford University School of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 80038
Record Dates: First submitted 2025-09-19; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants implanted with VNS (Other): Participants receiving vagus nerve stimulation through an implanted Vagus Nerve Stimulation Device.
  Interventions: Device: Vagus Nerve Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — Participants receiving vagus nerve stimulation through an implanted Vagus Nerve Stimulation Device.

SUMMARY:
The study will examine the autonomic, physiologic and neurophysiologic effects of implanted Vagus Nerve Stimulation (VNS) in treatment-resistant depression patients.

DETAILED DESCRIPTION:
The purpose of this study is to examine the autonomic and physiologic effects of implanted VNS in treatment-resistant depression patients. To examine the neurophysiologic effects of Vagus Nerve Stimulation (VNS) in treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years old.
2. Participants must be able to read, understand and have the capacity to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.
3. Proficiency in English sufficient to complete questionnaire and follow instructions during fMRI assessments and iTBS interventions.
4. Willingness to comply with all study procedures and the ability to communicate with study personnel about adverse events and other clinically important information
5. Participant must be currently enrolled in the REVEAL study and implanted with a VNS device for the clinical indication of Major Depressive Disorder (MDD)

   a. Clinical Indication of MDD as defined: Participant has a diagnosis of chronic (≥ 2 years) or ≥ 4 recurrent depressive episodes as defined by DSM-5 criteria documented using the MINI criteria and psychiatric medical record review.
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
7. Access to ongoing psychiatric care before and after completion of the study.
8. In good general health, as evidenced by medical history
9. Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

1. Participant is pregnant
2. Participant does not speak or read English
3. Any other clinical reasons deemed by the investigator of the study for which the participant would not be an appropriate candidate for the study.
4. Contraindication to MRI (ferromagnetic metal in their body)
5. Contraindication to EEG
6. Medication Contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gamma and theta band phase-amplitude coupling | Baseline, Week 6 and Week 19
  Measurement of EEG and ECG to quantify changes in phase-amplitude coupling in the gamma and theta band related to chronic VNS

SECONDARY OUTCOMES:
Resting state functional connectivity between the left dorsolateral prefrontal cortex and subgenual anterior cingulate cortex | Baseline, Week 6 and Week 19
  Measurement of changes in resting state functional connectivity between the left dorsolateral prefrontal cortex and subgenual anterior cingulate cortex with chronic VNS using fMRI.
Heart brain coupling | Week 19
  Measurement of heart brain coupling (heart rate entrainment in response to trains of intermittent theta burst stimulation) with VNS via an EKG sweep
Heart rate | Baseline, Week 6 and Week 19
  Measure heart rate and heart rate variability with VNS

OTHER OUTCOMES:
Galvanic Skin Response | Baseline, Week 6 and Week 19
  Measure the changes in sweat gland activity that affects the skin's electrical properties with VNS
Blood pressure | Baseline, Week 6 and Week 19
  Measure the changes in blood pressure with VNS
Respiratory rate | Baseline, Week 6 and Week 19
  Measure the changes in respiratory rate with chronic VNS.
Pupil diameter | Baseline, Week 6 and Week 19
  Measure the changes in pupil diameter with chronic VNS using pupillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Austelle, MD, Study Director — Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine